CLINICAL TRIAL: NCT01586000
Title: A Dose-finding Study to Evaluate the Effect of a Contraceptive Vaginal Ring, Releasing Nestorone® and Estradiol, on Cycle Control, Ovulation Inhibition, and Pharmacokinetics in Normal Cycling Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kimberly Myer (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Population Council (Other)
Responsible Party: Sponsor-Investigator, Kimberly Myer, Program Director, Premier Research
Organization: Premier Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCN012
Record Dates: First submitted 2012-03-19; First posted 2012-04-26 (Estimated); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2022-06

CONDITIONS: Suppression of Ovulation
Keywords: vaginal ring

ARMS (3):
- 10 µg/day E2 (Experimental): Two consecutive 3-month (90-day) rings will be used continuously for six months (180 days).
  Interventions: Drug: 10 µg/day E2 with NES 200® µg/day
- 20 µg/day E2 (Experimental): Two consecutive 3-month (90-day) rings will be used continuously for six months (180 days).
  Interventions: Drug: 20 µg/day E2 with NES 200® µg/day
- 40 µg/day E2 (Experimental): Two consecutive 3-month (90-day) rings will be used continuously for six months (180 days).
  Interventions: Drug: 40 µg/day E2 with NES 200® µg/day

INTERVENTIONS:
Drug: 10 µg/day E2 with NES 200® µg/day — 10 µg/day E2 with NES 200® µg/day delivered by CVR continuously for 6 months (180 days)
  Arms: 10 µg/day E2
Drug: 20 µg/day E2 with NES 200® µg/day — 20 µg/day E2 with NES 200® µg/day delivered by CVR continuously for 6 months (180 days)
  Arms: 20 µg/day E2
Drug: 40 µg/day E2 with NES 200® µg/day — 40 µg/day E2 with NES 200® µg/day delivered by CVR continuously for 6 months (180 days)
  Arms: 40 µg/day E2

SUMMARY:
This clinical trial is an experimental research study using a potential new form of birth control. Clinical trials include people who volunteer to take part in a study. Take your time to decide if you want to be part of this experimental research study. If you want to know more about this study first, ask the study doctor or study site staff. The investigators can also give you the study information written for doctors and clinic staff.

ELIGIBILITY:
Inclusion Criteria:

Women who meet all the following criteria are eligible for enrollment in the trial:

1. Healthy women of reproductive age (18-39 years, inclusive, at the enrollment visit).
2. Have a regular menstrual cycle that is 21-35 days in duration.
3. Have intact uterus and both ovaries.
4. Will be able and willing to comply with the protocol and sign an informed consent.
5. Will not be at risk for pregnancy. They will be consistently using a non-hormonal method, have a surgically sterile male partner with a vasectomy, be abstinent, or be in a same-sex relationship from the control period through study exit (including recovery period).
6. Will have diastolic blood pressure (BP) ≤85 mm Hg and systolic BP ≤135 mm Hg after 5 minutes in sitting position.
7. Willing to abstain from use of non-water based vaginal lubricant during the study.

Exclusion Criteria:

Women who meet any of the following criteria are not eligible for enrollment in the trial:

1. Participating in another clinical trial involving an investigational product within the last 30 days (prior to screening) or planning to participate in another clinical trial during this study.
2. Not living in the catchment area of the clinic.
3. Known hypersensitivity to progestins or estrogen.
4. All contraindications to combined estrogen-progestin contraceptive use including:

   * Thrombophlebitis or thromboembolic disorders.
   * Past personal history of deep vein thrombophlebitis or thromboembolic disorders.
   * History of venous thrombosis or embolism in a first-degree relative <55 years of age suggesting familial defect in blood coagulation system, which in the opinion of the investigator, suggests use of a hormonal contraceptive could pose a significant risk.
   * History of stroke.
   * Known or suspected carcinoma of the breast.
   * Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia.
   * Undiagnosed abnormal genital bleeding.
   * Cholestatic jaundice of pregnancy or jaundice with prior oral contraceptive use.
   * Hepatic adenomas or carcinomas.
   * Known or suspected pregnancy.
   * Smoking in women who are 35 years and over or will be 35 years during the course of the trial; women <35 years who smoke 15 cigarettes or more per day must be evaluated by the investigator for inclusion based on risk factors that would increase their risk for cardiovascular disease (CVD) and thromboembolism, e.g. lipid levels, glucose level, BP, BMI, family history of CVD at a young age.
   * History of retinal vascular lesions, unexplained partial or complete loss of vision.
   * Headaches with focal neurological symptoms (e.g., migraines with auras).
5. Desire to become pregnant during the study.
6. Breastfeeding.
7. Undiagnosed vaginal discharge or vaginal lesions or abnormalities. Subjects diagnosed at screening with a Chlamydia or gonococcus infection may be included in the trial following treatment; partner treatment is also recommended. Subjects with vaginitis (yeast, trichomonas, or bacterial vaginitis) may be enrolled after treatment. Investigators should make a determination if subjects are at high risk for reinfection, e.g. multiple sex partners, untreated partner, and whether such subjects can be included. In accordance with PI/medical designee assessment and local standards of practice, women with a history of genital herpes can be included if outbreaks are infrequent.
8. A clinically significant Pap test abnormality, as managed by current local or national guidelines. Women with a current abnormal Pap (within the last nine months):

   * In accordance with the Bethesda system of classification: smear suggestive of high-grade pre-cancerous lesion(s), including high grade squamous intraepithelial lesions (HGSILs), are excluded;

     * Women with low grade squamous intraepithelial lesion (LGSIL) or atypical squamous cells of undetermined significance (ASCUS)/high-risk human papillomavirus (HPV) positive, or Atypical squamous cells, cannot rule out a high grade lesion (ASC-H) may participate if further evaluated with colposcopy and biopsy determines no evidence of a lesion with a severity greater than cervical intraepithelial neoplasia (CIN) I.
     * Women with a biopsy finding of CIN I should have follow-up for this finding per standard of care; women are excluded if treatment is indicated.
   * In accordance with other Pap class systems:

     * Women with high grade dysplasia are excluded.
     * Women with low grade dysplasia or CIN I interpretation on Pap test may participate following exclusion of a high grade lesion by colposcopic evaluation based on Investigator discretion and provided there is appropriate follow up in accordance with local standards.
9. Known benign or malignant liver tumors; known active liver disease.
10. Invasive cancer (past history of any carcinoma or sarcoma, except non-melanoma skin cancer).
11. Current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive.
12. Known or suspected current alcoholism or drug abuse.
13. Elevated serum fasting clinical chemistry values or complete blood count (CBC) values designated clinically significant by the investigator or medically qualified sub-investigator.
14. Uncontrolled thyroid disease.
15. Known impaired hypothalamic-pituitary-adrenal reserve.
16. Body mass index (BMI) >35.
17. Use of injectable contraceptives (e.g. cyclofem or depo-medroxyprogesterone acetate) during the 6 months prior to enrollment or no spontaneous menses since last injection.
18. Use of oral contraceptives within one month prior to start of control cycle (subjects must undergo informed consent process and screening procedures before stopping oral contraceptives to participate in the study).
19. Use of hormonal contraceptives. NOTE: Removal of implanted hormonal contraceptives must have been for personal reasons unrelated to the purpose of enrollment in this study.
20. Current use of an intrauterine device (IUD). NOTE: Removal of an IUD must have been for personal reasons unrelated to the purpose of enrollment in this study.
21. Known hypersensitivity to silicone rubber.
22. History of toxic shock syndrome.
23. Cystoceles or rectoceles or other anatomical abnormality that would preclude use of a vaginal ring.
24. Planning to undergo major surgery during the study.
25. Severe constipation.
26. Use of liver enzyme inducers or inhibitors on a regular basis.
27. Known HIV infection.
28. Bariatric surgery within the past year prior to enrollment.
29. Any abnormalities found during the transvaginal ultrasound (TVUS) that the PI or medically qualified sub-investigator deems to put the subject at risk.
30. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - NYU School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Univeristy of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Started | 67 | 66 | 64
Completed | 45 | 47 | 47
Not Completed | 22 | 19 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 µg/Day E2 | 20 µg/Day E2 | 40 µg/Day E2 | Total
Number analyzed (Participants) | 67 | 66 | 64 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 67 | 66 | 64 | 197
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 28.8 [18 to 40] | 28.2 [18 to 38] | 29.6 [18 to 39] | 28.8 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 64 | 197
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 10 | 29
  Not Hispanic or Latino | 57 | 57 | 54 | 168
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 28 | 31 | 20 | 79
  White | 33 | 27 | 34 | 94
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7 | 14
Marital Status [Count of Participants; unit: Participants]
  Never Married | 50 | 41 | 43 | 134
  Married | 10 | 17 | 11 | 38
  Divorced | 5 | 4 | 8 | 17
  Separated | 2 | 2 | 2 | 6
  Widowed | 0 | 2 | 0 | 2
Highest Level of Education Completed [Count of Participants; unit: Participants]
  Has not completed high school | 0 | 1 | 2 | 3
  High school diploma or equivalent | 10 | 8 | 6 | 24
  Some college | 24 | 28 | 29 | 81
  College degree or higher | 33 | 29 | 27 | 89
Alcohol Use [Count of Participants; unit: Participants]
  Never | 8 | 7 | 13 | 28
  Former | 3 | 5 | 1 | 9
  Current | 56 | 54 | 50 | 160
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (4.210) | 25.35 (4.412) | 25.70 (4.232) | 25.82 (4.287)

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Bleeding is Reported.
Description: The primary outcome will be the number of days that bleeding or spotting is reported in the first 3 cycles (90 days) of treatment.
Time Frame: Three months
Population: All Safety population subjects with at least one non-missing bleeding record (from their diaries). All subjects enrolled in the study were included in the Safety population. In total, 2 subjects (both in the 200 µg/day NES and 40 µg/day E2 group) were not included in the Bleeding and Ovulation populations
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 67 | 66 | 62
Days
  Bleeding or Spotting | 34.0 (23.17) | 42.1 (24.51) | 39.8 (22.83)
  Bleeding Only | 14.7 (15.36) | 16.3 (16.3) | 15.0 (14.80)
  Spotting Only | 19.3 (18.61) | 25.8 (22.2) | 24.8 (19.06)

2. Secondary Outcome: Number of Subjects With Ovulation at During Each Cycle
Description: A subject will be considered to have ovulated if she has two consecutive progesterone values of ≥10 nmol/L (≥3 ng/mL) preceded by a follicular measurement of >10 mm in the previous 10 days. Number of subjects considered to have ovulated during each cycle is reported.
Time Frame: Control Cycle 1, Treatment Cycles 2, 3, and 7, Recovery Cycle 8, up to 8 months
Population: All Safety population subjects that had any cycle with a progesterone value and a TVUS assessment. All subjects enrolled in the study were included in the Safety population. In total, 2 subjects (both in the 200 µg/day NES and 40 µg/day E2 group) were not included in the Bleeding and Ovulation populations
Measure: Count of Participants; unit: Participants
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 67 | 66 | 62
Participants
  Control Cycle 1 | 0 | 2 | 0
  Treatment Cycle 2 | 27 | 25 | 25
  Treatment Cycle 3: number analyzed (Participants) | 60 | 60 | 59
  Treatment Cycle 3 | 21 | 19 | 20
  Treatment Cycle 7: number analyzed (Participants) | 46 | 48 | 47
  Treatment Cycle 7 | 18 | 15 | 14
  Recovery Cycle 8: number analyzed (Participants) | 57 | 56 | 53
  Recovery Cycle 8 | 7 | 2 | 3

3. Secondary Outcome: Area Under the Curve of NES and E2 at Specified Time Points
Description: Pharmacokinetic assessments will be performed to measure absorption in a substudy of 22 women (7-8 in each dose group) at a single center (Oregon Health and Science University) at initiation of each ring use and at final ring removal. Blood will be collected for measurements before insertion of the first ring (at Visit 12), before removal of the second ring (at Visit 41), and at 2, 4, 6, 8, 10, 12, 24, 48 and approximately 72 hours after the first ring is inserted (at Visit 12) and after the second ring is removed (at Visit 41). PK samples will also be collected at the time of removal of the first ring (0 hours) at Visit 32, 2 hours after removal of the first ring and insertion of the second ring, and at 24 hours after removal of the first ring and insertion of the second ring.
Time Frame: Visits 12, 32, and 41 (Treatment Period)
Population: The number analyzed at each time point is dependent on the number of subjects that completed each time point.
Measure: Mean (Standard Deviation); unit: hour*pg/mL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 7 | 7 | 8
hour*pg/mL
  Visit 12 NES 0-72 hrs post Ring 1 Insertion | 38685.7 (9770.06) | 31201.4 (4912.98) | 32845.0 (5370.53)
  Visit 32 NES 0-24 hrs after Removal of Ring 1 and Insertion of Ring 2: number analyzed (Participants) | 5 | 6 | 6
  Visit 32 NES 0-24 hrs after Removal of Ring 1 and Insertion of Ring 2 | 12906.4 (2574.38) | 16495.3 (3512.32) | 14073.3 (1729.37)
  Visit 41 NES 0-72 hrs post Ring 2 Removal: number analyzed (Participants) | 6 | 6 | 8
  Visit 41 NES 0-72 hrs post Ring 2 Removal | 742.7 (352.83) | 902.0 (460.43) | 863.5 (361.81)
  Visit 12 E2 0-72 hrs post Ring 1 Insertion: number analyzed (Participants) | 6 | 7 | 8
  Visit 12 E2 0-72 hrs post Ring 1 Insertion | 3690.77 (1414.324) | 4910.31 (1067.716) | 3648.83 (1341.309)
  Visit 32 E2 0-24 hrs after Removal of Ring 1 and Insertion of Ring 2: number analyzed (Participants) | 5 | 6 | 6
  Visit 32 E2 0-24 hrs after Removal of Ring 1 and Insertion of Ring 2 | 1237.10 (605.026) | 2470.0 (801.086) | 1198.83 (453.937)
  Visit 41 E2 0-72 hrs post Ring 2 Removal: number analyzed (Participants) | 5 | 6 | 8
  Visit 41 E2 0-72 hrs post Ring 2 Removal | 2098.36 (628.917) | 3208.62 (2470.399) | 2317.45 (963.316)

4. Secondary Outcome: The Safety of Administering 200 µg/Day of NES and One of Three Doses (10, 20, or 40 µg/Day) of E2 Delivered by CVR Continuously for 6 Months (180 Days).
Description: Clinical safety will be evaluated by collection of adverse events (AEs).
Time Frame: Through Recovery Cycle 8, up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 67 | 66 | 64
Participants
  Total Number of Subjects with at Least One AE | 58 | 57 | 55
  Total Number of Subjects with at Least One AE Leading to Discontinuation | 7 | 7 | 4
  Total Number of Subjects with at Least One Mild AE | 22 | 21 | 26
  Total Number of Subjects with at Least One Moderate AE | 34 | 32 | 26
  Total Number of Subjects with at Least One Severe AE | 2 | 4 | 3
  Total Number of Subjects with at Least One AE Probably Related | 11 | 9 | 5
  Total Number of Subjects with at Least One AE Highly Probably Related | 1 | 3 | 1
  Total Number of Subjects with at Least One SAE | 0 | 0 | 1

5. Secondary Outcome: Number of Days Bleeding is Reported.
Description: The primary outcome will be the number of days that bleeding or spotting is reported in the last 3 cycles (90 days) of treatment.
Time Frame: Three months
Population: All subjects enrolled in the study were included in the Safety population. In total, 2 subjects (both in the 200 µg/day NES and 40 µg/day E2 group) were not included in the Bleeding and Ovulation populations
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 67 | 66 | 62
Days
  Bleeding or Spotting | 31.3 (27.07) | 38.1 (31.12) | 30.8 (28.54)
  Bleeding Only | 8.2 (11.81) | 13.7 (22.89) | 8 (12.36)
  Spotting Only | 23.1 (23.19) | 24.4 (24.42) | 22.8 (25.1)

6. Secondary Outcome: Changes From Baseline in Albumin (g/dL)
Description: Clinical safety will also be evaluated by changes from baseline through end of treatment of blood chemistry and hematologic profile to assess safety of the three treatment groups.
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
g/dL | 0.01 (0.294) | -0.09 (0.281) | -0.02 (0.330)

7. Secondary Outcome: Changes From Baseline in ALT/SGPT (U/L)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
U/L | 2.6 (23.18) | -0.2 (7.72) | -1.4 (10.64)

8. Secondary Outcome: Changes From Baseline in AST/SGOT (U/L)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
U/L | 4.0 (43.51) | -2.7 (7.53) | -1.8 (16.57)

9. Secondary Outcome: Changes From Baseline in BUN (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
mg/dL | 0.5 (3.04) | 0.8 (3.45) | 1.0 (2.99)

10. Secondary Outcome: Changes From Baseline in Calcium (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
mg/dL | -0.02 (0.434) | -0.16 (0.434) | 0.00 (0.447)

11. Secondary Outcome: Changes From Baseline in Creatinine (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
mg/dL | 0.035 (0.1116) | 0.041 (0.0969) | 0.046 (0.0827)

12. Secondary Outcome: Changes From Baseline in Glucose (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
mg/dL | 2.2 (13.61) | 2.7 (11.97) | 1.5 (14.20)

13. Secondary Outcome: Changes From Baseline in GGT (U/L)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 55 | 58 | 53
U/L | 1.0 (5.67) | 2.5 (5.56) | 2.1 (7.67)

14. Secondary Outcome: Changes From Baseline in Total Bilirubin (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
mg/dL | -0.03 (0.212) | -0.07 (0.227) | -0.03 (0.227)

15. Secondary Outcome: Changes From Baseline in Total Protein (g/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
g/dL | 0.00 (0.488) | -0.11 (0.455) | -0.03 (0.468)

16. Secondary Outcome: Changes From Baseline in Total Cholesterol (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 60 | 56
mg/dL | -6.6 (23.26) | -9.5 (23.79) | -37.9 (24.83)

17. Secondary Outcome: Changes From Baseline in HDL Cholesterol (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 60 | 56
mg/dL | -3.9 (11.70) | -7.0 (10.84) | -3.5 (11.86)

18. Secondary Outcome: Changes From Baseline in LDL Cholesterol (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 60 | 56
mg/dL | -5.3 (24.05) | -4.8 (25.01) | -7.8 (21.54)

19. Secondary Outcome: Changes From Baseline in Triglycerides (mg/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 60 | 56
mg/dL | 0.2 (34.05) | 0.4 (31.81) | 4.6 (40.70)

20. Secondary Outcome: Changes From Baseline in Chloride (mmol/L)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
mmol/L | 1.5 (2.75) | 2.3 (2.09) | 1.2 (3.00)

21. Secondary Outcome: Changes From Baseline in Potassium (mmol/L)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
mmol/L | -0.11 (0.446) | -0.12 (0.414) | -0.14 (0.456)

22. Secondary Outcome: Changes From Baseline in Sodium (mmol/L)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 57
mmol/L | 0.6 (2.72) | 1.3 (2.83) | 0.3 (2.70)

23. Secondary Outcome: Changes From Baseline in RBC (MIL/uL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: MIL/uL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 56 | 62 | 58
MIL/uL | -0.004 (0.2342) | -0.062 (0.2260) | 0.032 (0.2855)

24. Secondary Outcome: Changes From Baseline in WBC (THOU/uL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: THOU/uL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 56 | 62 | 58
THOU/uL | 0.028 (1.4519) | 67.522 (532.9508) | 0.089 (1.8263)

25. Secondary Outcome: Changes From Baseline in Hemoglobin (g/dL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 57 | 62 | 58
g/dL | -0.21 (0.772) | -0.38 (0.798) | -0.25 (0.950)

26. Secondary Outcome: Changes From Baseline in Hematocrit (%)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 56 | 62 | 58
percentage | -0.41 (2.337) | -0.99 (2.269) | -0.45 (2.770)

27. Secondary Outcome: Changes From Baseline in Platelet Count (THOU/uL)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: THOU/uL
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 56 | 62 | 58
THOU/uL | -3.0 (45.50) | 4.6 (29.92) | 20.8 (32.88)

28. Secondary Outcome: Changes From Baseline in Basophils (%)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 54 | 57 | 55
percentage | 3.19 (16.656) | 0.20 (0.524) | -0.52 (4.283)

29. Secondary Outcome: Changes From Baseline in Eosinophils (%)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 54 | 57 | 56
percentage | -0.180 (5.1571) | 0.198 (1.8886) | -1.054 (8.2595)

30. Secondary Outcome: Changes From Baseline in Lymphocytes (%)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 54 | 57 | 56
percentage | -0.141 (13.1510) | 2.919 (10.7313) | 2.518 (12.7415)

31. Secondary Outcome: Changes From Baseline in Monocytes (%)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 54 | 57 | 56
percentage | -0.310 (3.2383) | -0.260 (4.9032) | 0.030 (3.4508)

32. Secondary Outcome: Changes From Baseline in Neutrophils (%)
Description: as for outcome 6
Time Frame: Visit 41 (end of Treatment Cycle 7) compared to Visit 1 (Screening)
Population: Change from Baseline to Final Evaluation. Subjects that had lab values at Visit 1 and Visit 41 were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
Number analyzed (Participants) | 54 | 55 | 55
percentage | 0.080 (18.6460) | 0.357 (19.6337) | -2.740 (22.3667)

ADVERSE EVENTS:
Time Frame: from enrollment through Recovery Cycle 8, up to 8 months
Arm/Group | 10 µg/day E2 | 20 µg/day E2 | 40 µg/day E2
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/66 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/66 | 1/64
Other Adverse Events (participants affected / at risk) | 58/67 | 57/66 | 55/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 µg/day E2 (N=67) | 20 µg/day E2 (N=66) | 40 µg/day E2 (N=64)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 µg/day E2 (N=67) | 20 µg/day E2 (N=66) | 40 µg/day E2 (N=64)
Headache (Nervous system disorders) | 28 (62) | 20 (62) | 14 (62)
Upper Respiratory Tract Infection (Infections and infestations) | 16 (43) | 13 (43) | 14 (43)
NASOPHARYNGITIS (Infections and infestations) | 9 (37) | 16 (37) | 12 (37)
Nausea (Gastrointestinal disorders) | 5 (25) | 10 (25) | 10 (25)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 (23) | 7 (23) | 6 (23)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 7 (22) | 10 (22) | 5 (22)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (19) | 5 (19) | 9 (19)
VAGINITIS BACTERIAL (Infections and infestations) | 8 (17) | 4 (17) | 5 (17)
DIARRHOEA (Gastrointestinal disorders) | 6 (16) | 4 (16) | 6 (16)
INFLUENZA (Infections and infestations) | 9 (16) | 5 (16) | 2 (16)
ACNE (Skin and subcutaneous tissue disorders) | 8 (15) | 6 (15) | 1 (15)
MOOD SWINGS (Psychiatric disorders) | 4 (14) | 7 (14) | 3 (14)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (12) | 4 (12) | 4 (12)
DIZZINESS (Nervous system disorders) | 3 (12) | 5 (12) | 4 (12)
FUNGAL INFECTION (Infections and infestations) | 3 (12) | 6 (12) | 3 (12)
ANXIETY (Psychiatric disorders) | 4 (11) | 3 (11) | 4 (11)
DYSPAREUNIA (Psychiatric disorders) | 4 (11) | 5 (11) | 2 (11)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (11) | 4 (11) | 4 (11)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 5 (11) | 2 (11) | 4 (11)
VOMITING (Gastrointestinal disorders) | 2 (10) | 4 (10) | 4 (10)
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 2 (10) | 4 (10) | 4 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No